CLINICAL TRIAL: NCT05192044
Title: Less Than 100 Hours Hospital Stay After Pancreatico-duodenectomy, RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Debakey4
Record Dates: First submitted 2021-12-30; First posted 2022-01-14 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-12

CONDITIONS: Pancreas Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Fast track Care (Enhanced recovery after)pancreatico-duodenectomy
  Interventions: Other: Fast track Care pancreatico-duodenectomy.
- Group B (Active Comparator): Conventional Care pancreatico-duodenectomy.
  Interventions: Other: Conventional Care

INTERVENTIONS:
Other: Fast track Care pancreatico-duodenectomy. — Enhanced recovery after pancreatico-duodenectomy, with early oral intake, mobilization & discharge
  Arms: Group A
Other: Conventional Care — Conventional Care
  Arms: Group B

SUMMARY:
Few decades back pancreatico-duodenectomy (PD) was associated with a very high morbidity and mortality. With recent advancements in surgical and anesthetic techniques and improvement in peri-operative care, PD has evolved into a procedure with acceptable morbidity and mortality. Today PD is associated with a mortality of less than 5%, in high volume tertiary care centers. The multimodal concept of fast-track surgery was first introduced in colonic surgery. Several studies have demonstrated the effectiveness of this program in colonic resection. Recently, fast-track surgery has been attempted in pancreatic surgery with encouraging results, but such data are sparse. The core aims of ERAS protocols are to safely hasten postoperative recovery and ease the stress response.

Specifically, in the context of pancreatico-duodenectomy, such interventions have been shown to be safe with no increase in mortality or unplanned readmissions, delayed gastric emptying (DGE), or pancreatic fistula . Purported benefits include reduced admission related costs, incidence of DGE, overall morbidity and length of stay.

The aim of this study was to evaluate the feasibility of implementing fast track rehabilitation protocol following pancreaticoduodenectomy and to see if it is associated with improved recovery, reduced morbidity and reduced length of hospital stay.

DETAILED DESCRIPTION:
Study population: This is a prospective study that will be conducted on all patients of both sexes and definite age groups attending the National Cancer Institute, Cairo University and candidate for pancreatico-duodenectomy Sampling: all cases fulfilling the inclusion criteria will be included in the study.

Patients will be classified into two groups:

* Group A: Fast track Care pancreatico-duodenectomy.
* Group B: Conventional Care pancreatico-duodenectomy. Baseline demographics, body mass index (BMI), perioperative parameters, postoperative course, postoperative complications and 30-days operative mortality will be analyzed.

Inclusion criteria:

* Age ≤ 75 years
* ASA 1 or 2
* BMI < 35 The underlying pathology or use of neoadjuvant chemotherapy did not preclude inclusion into the study

Exclusion criteria:

* pancreatico-duodenectomy with vascular reconstruction.
* Unenthusiastic patients.

Type of study: randomized controlled trial The assignment of patients to either group will be done by a random computer-assissted allocation. The allocation will be done by the use of opaque envelopes with assignments.

It's an open-labeled study i.e. patients, investigators (surgeons, researchers) and data collectors will know which procedure will be done to which patients.

Discharge criteria for goup A include; uncomplicated procedure, afebrile patient without tachycardia, tolerance of oral feeding, adequate control of pain with oral analgesia, patient ambulating independently, adequate support at home.

Follow up: will be completed within one month (immediate post-operative outcome).

ELIGIBILITY:
Inclusion Criteria:

* Age ≤ 75 years
* ASA 1 or 2
* BMI < 35
* The underlying pathology or use of neoadjuvant chemotherapy did not preclude inclusion into the study

Exclusion Criteria:

- pancreatico-duodenectomy with vascular reconstruction.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-12-25 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of enhanced recovery after pancreatico-dudenectomy | 1 month after surgery
  Feasibility will be measured by recording post operative complications according to Clavien- Dindo classification

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Mahmoud, Professor, Study Director — National Cancer Institute, Cairo University, Egypt
Locations (1):
- National Cancer Institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
In a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After publication & for a year
Access Criteria: The journal of publication